CLINICAL TRIAL: NCT06964711
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Dose and Multiple Ascending Dose, Single Center Phase1 Study of Safety, Tolerability and Pharmacokinetics of GW117 ODT in Healthy Volunteers
Brief Title: GW117 ODT （Orally Disintegrating Tablets） Safety and Pharmacokinetics Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Greatway Pharmaceutical Technology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW117-C102; CTR20221750 (Other: Chinadrugtrials Number)
Record Dates: First submitted 2025-04-22; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: MDD; GW117; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GW117 ODT (Orally disintegrating tablet) (Experimental): Take the tablet sublingually, Once daily SAD: Take once only，0.5mg，1mg，2mg，4mg MAD: Take for 7 consecutive days，1mg，2mg
  Interventions: Drug: GW117 ODT
- Placebo (Placebo Comparator): Take the tablet sublingually, Once daily SAD: Take once only MAD: Take for 7 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW117 ODT — Sublingual route ， 0.5mg/1mg/2mg/4mg，QD
  Other Names: GW117 Orally Disintegrating Tablets
  Arms: GW117 ODT (Orally disintegrating tablet)
Drug: Placebo — GW117 Placebo matching for Sublingual route ，QD
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetics of single and multiple ascending doses of GW117 ODT in healthy volunteers

DETAILED DESCRIPTION:
Single ascending dose (SAD), multiple ascending dose (MAD), double-blind placebo-controlled study in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body weight should be at least 50.0kg for males and 45.0kg for females, with body mass index (weight/height 2) in the range of 19-26 kg/m2
* The results of physical examination were normal or abnormal without clinical significance;
* The results of vital signs were normal or abnormal without clinical significance
* The results of laboratory tests (blood routine, urine routine, liver function, renal function, blood glucose, electrolytes, coagulation function) were normal or abnormal without clinical significance
* negative results of pregnancy examination
* normal serological test results (five hepatitis B tests, hepatitis C antibodies, syphilis sero-specific antibodies, HIV antibodies)
* Normal or approximately normal or abnormal results of 12-lead electrocardiogram were not clinically significant
* Normal or abnormal chest X-ray findings had no clinical significance
* The normal or abnormal results of abdominal ultrasound had no clinical significance;
* Alcohol breath test results were negative
* Urine nicotine test results were negative
* Urine drug screening (morphine, methamphetamines, ketamine, dimethylenedioxyamphetamine, and tetrahydrocannabinol acid) was negative

Exclusion Criteria:

* Allergic constitution or a history of drug or food allergy
* any medical history that may affect the safety of the trial or the in vivo course of the drug
* any history of surgery or trauma that may affect the safety of the trial or the course of the drug in vivo
* currently suffering from any unstable or recurrent disease or disease affecting the course of the drug in vivo
* a history of drug abuse/dependence in the past 2 years
* any medications used within 14 days before the test
* smoking within 2 weeks before medication or during the study period;
* alcohol abuse [drinking more than 14 units of alcohol per week in the 3 months before screening (1 unit of alcohol ≈360mL of 5% beer or 45mL of 40% spirits or 150mL of 12% wine)], or drinking alcohol within 1 week before medication, or unable to abstain from alcohol during the study
* participated in other drug clinical trials within 90 days before the trial
* blood loss or donation of 400mL or more within 90 days before the test;
* a history of fainting or bleeding
* lactating women
* plan to donate sperm or egg, plan to have children, or be unwilling or unable to take effective contraceptive measures within 30 days before the trial to 6 months after the end of the trial
* abnormal neurological or mental status or language disorder
* patients with abnormal saliva secretion, severe oral ulcer or other oral mucosal diseases;
* The investigators considered that they were not suitable to participate in the trial due to other circumstances

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with at least one safety event | baseline up to Day 9
  Safety will be evaluated by the monitoring of adverse events (AEs), vital signs, electrocardiogram (ECG) evaluations, clinical laboratory assessments, and physical examination findings.
  Percentage of participants who experience at least one treatment-emergent adverse event (TEAE) will be captured.

SECONDARY OUTCOMES:
Pharmacokinetics -maximum plasma concentration (Cmax) | baseline up to Day 8
  Determination of maximum plasma concentration (Cmax)
Pharmacokinetics - time to maximum concentration (Tmax) | baseline up to Day 8
  Determination of time to maximum concentration
Pharmacokinetics - plasma exposure (AUC0-t, AUC0-inf) | baseline up to Day 8
  Determination of plasma exposure (AUC0-t, AUC0-inf)
Pharmacokinetics - terminal elimination half life (t1/2) | baseline up to Day 8
  Determination of terminal half life

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No